CLINICAL TRIAL: NCT06205199
Title: Analgesic Effect of Ropivacaine Hydrochloride Combined With Hydromorphone Hydrochloride for Combined Spinal-epidural Anesthesia After Total Knee Arthroplasty
Brief Title: Analgesic Effect of Ropivacaine Combined With Hydromorphone for CSEA After Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2ed hosp JLU ana dept
Record Dates: First submitted 2023-12-17; First posted 2024-01-12 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Postoperative Analgesia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: The participants, the surgeon, the surgical nurse, the data collector, and the anesthesiologist administering anesthesia were not aware of the patient groups
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydromorphone group (Experimental): Hydromorphone 50 micrograms combined with ropivacaine 15 mg was injected into the subarachnoid space
  Interventions: Drug: Hydromorphone was injected into the subarachnoid space
- Control group (No Intervention): Ropivacaine 15 mg was injected into the subarachnoid space

INTERVENTIONS:
Drug: Hydromorphone was injected into the subarachnoid space — The dose of hydromorphone is 50 micrograms
  Arms: Hydromorphone group

SUMMARY:
The aim of this study is to investigate the continuous analgesic effect and side effects of ropivacaine combined with hydromorphone for combined spinal-epidural anesthesia(CSEA) after total knee arthroplasty and to explore its clinical application value. To observe whether hydromorphone combined with ropivacaine can promote the rapid recovery of patients.

DETAILED DESCRIPTION:
For patients undergoing total knee arthroplasty, different spinal anesthesia drugs were injected in the two groups. The spinal anesthetic drugs injected in the hydromorphone group were hydromorphone 50 μg and ropivacaine 15 mg. In the control group, the spinal anesthetic was ropivacaine 15 mg.The differences in analgesia, sedation, and side effects between the hydromorphone group and the control group were analyzed by collecting various data at different times after anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Age between 55 and 80 years old.
* ASA grade I to III.
* BMI:20-29kg/m2.
* No recent use of sedatives, opioids, or other analgesics.
* There was no contraindication of spinal anesthesia, severe dysfunction of heart, lung and other important organs or serious systemic diseases.
* Patients were willing to participate in the study and signed the informed consent.

Exclusion Criteria:

* The patient has mental illness or cannot cooperate with the completion of spinal anesthesia.
* The patient had a history of spinal surgery and spinal deformity.
* Patients had a history of opioid intolerance or adverse reactions.
* puncture site infection, coagulopathy or recent use of anticoagulant drugs.
* History of allergy to local anesthetics.
* Failed puncture.
* Unable to cooperate to complete the research process.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2022-10-27 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Incidence of moderate to severe pain at rest at 6, 12, 18, and 24 hours after anesthesia. | 6, 12, 18, and 24 hours after anesthesia
  The NRS scale was used to evaluate pain scores at rest at 6, 12, 18, and 24 hours after anesthesia；Numeric rating scale (NRS, an 11-point scale where 0=no pain and 10=worst possible pain)
Incidence of moderate to severe pain with movement at 6, 12, 18, and 24 hours after anesthesia. | 6, 12, 18, and 24 hours after anesthesia
  NRS rating scale was used to evaluate pain score during movement at 6 hours, 12 hours, 18 hours, and 24 hours after anesthesia；Numeric rating scale (NRS, an 11-point scale where 0=no pain and 10=worst possible pain)

SECONDARY OUTCOMES:
Sedation and agitation at 6, 12, 18 and 24 hours after anesthesia | 6, 12, 18, and 24 hours after anesthesia
  RASS was used to assess sedation and agitation at 6, 12, 18, and 24 hours after anesthesia；Richmond Agitation and Sedation Scale(RASS,a 10-point scale where -5=unwakeable,0=clear and calm,+4=aggressive)
The number of effective compressions of PCIA at 24 hours after surgery | Postoperative 24 hours
  Effective number of PCIA compressions during the 24 hours after surgery
The proportion of the required additional analgesia after 24 hours | Postoperative 24 hours
  The proportion of patients requiring additional analgesia 24 hours after surgery in the whole group
Total non-steroidal analgesic drug consumption 48 hours after surgery | Postoperative 48 hours
  Non-steroidal analgesic consumption at 48 hours after surgery
Total opioid analgesic consumption at 48 hours after surgery | Postoperative 48 hours
  Opioid analgesic consumption at 48 hours after surgery
The proportion of getting out of bed within 48h | Postoperative 48 hours
  The proportion of people who got out of bed 48 hours after operation in the whole group
Satisfaction with postoperative analgesia | 5 days after surgery
  Patient satisfaction with postoperative analgesia；0=unsatisfied, 10=fully satisfied
Retention time of urinary tube | 5 days after surgery
  Retention time of urinary catheter after surgery
Length of postoperative hospital stay | 2 weeks after surgery
  The hospitalization days after surgery
The incidence of postoperative nausea or vomiting | Postoperative 48 hours
  Nausea and vomiting accounted for the proportion of the whole group
The incidence of postoperative pruritus | Postoperative 48 hours
  Pruritus accounted for the proportion of the whole group
The incidence of intraoperative hypotension | During the operation
  Systolic blood pressure drops to 20% of basal blood pressure or systolic blood pressure drops below 90mmHg
The incidence of intraoperative hypoxemia | During the operation
  SpO2 drop below 90%
Incidence of intraoperative HR reduction | During the operation
  HR < 45 beats /min

CONTACTS AND LOCATIONS:
Overall Officials: Dan Tian, Principal Investigator — Second Hospital of Jilin University
Locations (1):
- Second Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No